CLINICAL TRIAL: NCT02898402
Title: Study on Seroprevalence and Risk Factors of Coxiella Burnetii (Q Fever) in the South of Reunion Island
Acronym: E-Q-RUN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/CHU/04
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: q Fever
MeSH Terms: conditions — Q Fever | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: blood sample and questionnaire — In addition to normal blood sample performed at entry before delivery, an extra 5 ml blood sample will be taken to establish Q fever serodiagnosis and a short questionnaire will be filled in for clinical and epidemiological data.

SUMMARY:
Emergent and infectious diseases are a public health priority on Reunion Island. Amongst public health threats, the infection due to Coxiella burnetii (Q fever) seems to have appeared on Reunion island in 2007 with two hospitalised confirmed cases (one death) and one probable case with a goat farmer.

According to the investigator, the diffusion of C. burnetti is more ancient and such diagnosis have been made in the last 30 years with 80 positive serologies identified between 2005 and 2011.

Considering the high epidemic power of this disease, its often silent clinical expression and its life-threatening condition, the principal investigator wishes to perform a sero-epidemiological study in order to establish or to reject the risk of emergence of Q fever in Reunion island.

The study will be performed on pregnant women because Q fever is responsible for particular complications during pregnancy and because the number of pregnancy followed on Reunion island is stable from one year to the other. The pregnant women population presenting the same exposure criteria as the general population, this population will be used to extrapolate to the general population of the island.

ELIGIBILITY:
Inclusion Criteria:

* all pregnant women coming to the two maternity hospitals located in the south of Reunion island during inclusion period who have been informed and gave consent to participate to the study.

Exclusion Criteria:

* women aged less than 18 years old.
* women who did not give their consent
* women for whom it is not possible to perform the blood sample.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pregnant women coming to hospital for delivery
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
prevalence of Coxiella burnetii infection in general population in the south of Reunion island | at inclusion
  Q fever seroprevalence obtained from blood samples taken on pregnant women hospitalised for delivery will be used to extrapolate to Reunion island general population Q fever seroprevalence.

IPD SHARING:
Plan to Share IPD: No